CLINICAL TRIAL: NCT04162223
Title: Mechanisms of Immunosenescence: A Single-Blinded Comparison of the Location of Vaccine Inoculum, Intramuscular Versus Subcutaneous Adipose Tissue, on the Immune Response of Healthy Elderly Adults to a Recombinant Hepatitis B Surface Antigen Vaccine (Recombivax-HB)
Brief Title: Hepatitis B Vaccine in Seniors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Marcelo Sztein, Professor of Pediatrics and Medicine, Microbiology and Immunology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0199221
Record Dates: First submitted 2019-10-31; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis B Vaccination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subcutaneous Fat Vaccine Injection (Experimental): Subcutaneous fat Hepatitis B vaccine injections on Days 0, 28, and 180.
  Interventions: Biological: Subcutaneous fat injection of Recombivax-HB
- Intramuscular Vaccine Injection (Experimental): Intramuscular Hepatitis B vaccine injections on Days 0, 28, and 180.
  Interventions: Biological: Intramuscular injection of Recombivax-HB

INTERVENTIONS:
Biological: Subcutaneous fat injection of Recombivax-HB — Subcutaneous fat injection administration of licensed Hepatitis B Surface Antigen Vaccine (Recombivax-HB) on Days 0, 28, and 180.
  Arms: Subcutaneous Fat Vaccine Injection
Biological: Intramuscular injection of Recombivax-HB — Intramuscular injection administration of licensed Hepatitis B Surface Antigen Vaccine (Recombivax-HB) on Days 0, 28, and 180.
  Arms: Intramuscular Vaccine Injection

SUMMARY:
The first purpose of this study is to test the body's protective reaction (making antibodies) to a licensed hepatitis B vaccine (Recombivax-HB) after it is injected either in the arm fat or muscle. Hepatitis B virus is an important cause of liver disease in humans. More than 21% of healthy adults over age 60 years demonstrate evidence of previous Hepatitis B infection using a common blood test.

The second purpose of this study is to learn more information about other reasons (such as body fat content, gene types, etc.), why older people respond less well than younger people to vaccines. The Investigators will also learn more about the ability of certain white blood cells, called T cells, to respond to protein signals in the blood. T cells do not seem to respond as well to these protein signals as individuals age. The Investigators will compare results to a younger group of volunteers who have also been vaccinated with hepatitis B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, community-dwelling adult men or women 65 years of age or older, of any race or ethnic group
* Medical history with stable chronic non-immunologically mediated medical conditions (e.g. osteoarthritis, hypertension)
* Normal (within the normal range for reference laboratory or clinically insignificant values as determined by the Principal Investigator) TSH, serum vitamin B12, AST/SGOT, ALT/SGPT
* Negative serum tests for hepatitis B surface antigen and antibody, hepatitis B core antibody and hepatitis C antibody
* Has given informed consent
* Ready access to a telephone

Exclusion Criteria:

* Clinically apparent or history of immunologically mediated diseases (e.g. rheumatoid arthritis, lupus erythematosis, etc.), immunodeficiency, severe cardiovascular disease, severe respiratory disease (requiring supplemental oxygen), endocrine disorder (e.g. thyroid dysfunction, adrenal insufficiency), liver disease (cirrhosis), renal disease, gastrointestinal disease, neurologic illness, psychiatric disorder (eligible if treated and in remission), drug or alcohol abuse or currently smoking 10 cigarettes per day
* Infections within 2 weeks of immunization (the most frequent infections are respiratory and urogenital)
* Inflammatory processes such as known chronic infections, inflammatory bowel disease or Westergren sedimentation rate (greater than 50mm/hour for men, greater than 60mm/hour for women)
* All malignancies (excluding non-melanotic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years
* Arteriosclerotic event during the 2 weeks prior to enrollment (e.g. medically documented myocardial infarction, stroke, recanalization of the femoral arteries, claudication, or Transient Ischemic Attack (TIA))
* Cardiac insufficiency, if heart failure present (New York Heart Association functional class III or IV)
* Poorly controlled hypertension (Systolic Blood Pressure 180mmHg, Diastolic Blood Pressure 100mmHg on two separate determinations at least 10 minutes apart)
* Renal Insufficiency (serum creatinine 2.0 or BUN 40) and stable over past 6 months
* Elevated or low glucose (fasting 140 or less than 70, non-fasting 200)
* Cognitive impairment: score of less than 23 on the Folstein Mini-Mental State Examination
* Depression or mood alteration: score of 6 on the Geriatric Depression Scale
* Malnutrition as defined by clinical judgment and by decreased serum albumin (less than 3.2g/L) or hypocholesterolemia (less than 160mg/dL), or low total lymphocyte count (less than 1500/ml3)
* Anemia (Hct less than 30% or low serum vitamin B12 or vitamin E level)
* History of or current alcoholism or consuming greater than 2oz of ETOH/day; current drug abuse; currently smoking 10 cigarettes per day
* Risk factors for hepatitis B (which would indicate the need for immediate immunization with licensed vaccine), such as parenteral drug abuse, multiple sexual partners, commercial sex worker, health care worker
* History of hepatitis B infection or vaccination
* Positive test for hepatitis B surface antigen or antibody, hepatitis B core antibody, or hepatitis C antibody
* History of significant bilateral upper arm injury or surgery, of any duration, because theoretically this may impede lymph drainage to regional lymph nodes
* Reported allergy to thimerosal (i.e., contact lens solution) or yeast products
* Unable to attend the Baltimore VA Medical Center or the Waxter Center on a regular basis; no telephone in primary residence
* Subcutaneous fat pad less than 6 mm in thickness as determined by computer tomography
* Medication exclusions include prednisone greater than 5 mg/day (or equal), colchicines, imuran, methotrexate, azathioprine, cyclophosphamide, cyclosporine, or interferons

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2000-03-29 (Actual); Primary Completion 2003-05-20 (Actual); Study Completion 2003-05-20 (Actual)

PRIMARY OUTCOMES:
Hepatitis B surface antibody (HBsAb) titers (in international units/L) | two years
  Basic science - Primary and booster hepatitis B surface antibody titers to three injections of Recombivax-HB in the elderly and young adults immunized subcutaneously or intramuscularly, including % responders
Cell-mediated immune responses (CMI) (levels of interferon gamma and other cytokines in pg/ml) | two years
  Basic science - Primary and booster CMI responses to three injections of Recombivax-HB in the elderly and young adults immunized subcutaneously or intramuscularly, including % responders

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Edelman R, Deming ME, Toapanta FR, Heuser MD, Chrisley L, Barnes RS, Wasserman SS, Blackwelder WC, Handwerger BS, Pasetti M, Siddiqui KM, Sztein MB. The SENIEUR protocol and the efficacy of hepatitis B vaccination in healthy elderly persons by age, gender, and vaccine route. Immun Ageing. 2020 Apr 28;17:9. doi: 10.1186/s12979-020-00179-9. eCollection 2020. PMID 32355503